CLINICAL TRIAL: NCT03269760
Title: Advancing the Multimodal Pathway: Investigating the Use of Sleep and Zolpidem in the Recovery After Shoulder Arthroplasty
Brief Title: Multimodal Sleep Pathway for Shoulder Arthroplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-20346
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Sleep Disturbance; Shoulder Arthritis; Arthroplasty Complications; Perioperative/Postoperative Complications
MeSH Terms: conditions — Parasomnias; Postoperative Complications | interventions — Zolpidem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention): Current practice of postoperative care without sleep medicine measures
- Interventional Sleep Medicine (Experimental): Use of a multimodal sleep pathway including non-pharmacological sleep hygiene interventions and the use of zolpidem to improve patient sleep, pain control, and subsequent recovery after undergoing total shoulder arthroplasty.
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Drug: Zolpidem — Addition of both non-pharmacologic nursing directed sleeping hygiene practices with pharmacologic zolpidem to improve sleep latency
  Other Names: Nursing sleep medicine protocol
  Arms: Interventional Sleep Medicine

SUMMARY:
The purpose of the study is to investigate the efficacy of sleep medicine in the recovery of orthopaedic shoulder arthroplasty patients. The investigators hypothesize that a multimodal sleep pathway including non-pharmacological sleep hygiene interventions and the use of zolpidem can improve patient sleep, pain control, and subsequent recovery after undergoing total shoulder arthroplasty.

DETAILED DESCRIPTION:
Shoulder pain at night is a common symptom of shoulder arthritis and contributes to sleep disturbances. Many patients also have difficulty sleeping after shoulder surgery due to the constraints of sling immobilization. While in the hospital, sleep is also disrupted due to pain, nursing staff, other patients, and bathroom use. While poor sleep may appear trivial, sleep deprivation in animal models has identified significant adverse effects on bone metabolism, bone mass, and recovery from post surgical pain.

Recent evidence has shown that non-pharmacological sleep interventions that improve sleep hygiene and duration can optimize athletic peak performance, fatigue, and recovery. Furthermore, pharmacological sleep aid use with zolpidem in orthopaedic postoperative patients has suggested safe administration, improved pain control, reduced pain medication use, and higher patient satisfaction in the settings of total knee and hip arthroplasty, rotator cuff repairs, and ACL reconstruction.

The purpose of the study is to investigate the efficacy of sleep medicine in the recovery of orthopaedic shoulder arthroplasty patients. The investigators hypothesize that a multimodal sleep pathway including non-pharmacological sleep hygiene interventions and the use of zolpidem can improve patient sleep, pain control, and subsequent recovery after undergoing total shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

All consenting adults undergoing elective total shoulder replacement

-

Exclusion Criteria:

* Allergies to zolpidem or refusal to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Lead's Sleep scale | postoperative day 1
  Patient reported outcome

SECONDARY OUTCOMES:
Sleep journals | postoperative day 1-7
  patient reported outcome
Pain scores | postoperative day 1
  ]pain scores

CONTACTS AND LOCATIONS:
Locations (1):
- Ucsf, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho CH, Lee SW, Lee YK, Shin HK, Hwang I. Effect of a sleep aid in analgesia after arthroscopic rotator cuff repair. Yonsei Med J. 2015 May;56(3):772-7. doi: 10.3349/ymj.2015.56.3.772. PMID 25837184
- [Background] Chouchou F, Khoury S, Chauny JM, Denis R, Lavigne GJ. Postoperative sleep disruptions: a potential catalyst of acute pain? Sleep Med Rev. 2014 Jun;18(3):273-82. doi: 10.1016/j.smrv.2013.07.002. Epub 2013 Sep 24. PMID 24074687
- [Background] Dolan R, Huh J, Tiwari N, Sproat T, Camilleri-Brennan J. A prospective analysis of sleep deprivation and disturbance in surgical patients. Ann Med Surg (Lond). 2016 Jan 6;6:1-5. doi: 10.1016/j.amsu.2015.12.046. eCollection 2016 Mar. PMID 26909151
- [Background] Gong L, Wang Z, Fan D. Sleep Quality Effects Recovery After Total Knee Arthroplasty (TKA)--A Randomized, Double-Blind, Controlled Study. J Arthroplasty. 2015 Nov;30(11):1897-901. doi: 10.1016/j.arth.2015.02.020. Epub 2015 Feb 24. PMID 26344094
- [Background] Krenk L, Jennum P, Kehlet H. Postoperative sleep disturbances after zolpidem treatment in fast-track hip and knee replacement. J Clin Sleep Med. 2014 Mar 15;10(3):321-6. doi: 10.5664/jcsm.3540. PMID 24634631
- [Background] Krenk L, Jennum P, Kehlet H. Sleep disturbances after fast-track hip and knee arthroplasty. Br J Anaesth. 2012 Nov;109(5):769-75. doi: 10.1093/bja/aes252. Epub 2012 Jul 24. PMID 22831887
- [Background] Mah CD, Mah KE, Kezirian EJ, Dement WC. The effects of sleep extension on the athletic performance of collegiate basketball players. Sleep. 2011 Jul 1;34(7):943-50. doi: 10.5665/SLEEP.1132. PMID 21731144
- [Background] Mulligan EP, Brunette M, Shirley Z, Khazzam M. Sleep quality and nocturnal pain in patients with shoulder disorders. J Shoulder Elbow Surg. 2015 Sep;24(9):1452-7. doi: 10.1016/j.jse.2015.02.013. Epub 2015 Apr 1. PMID 25842028
- [Background] Tompkins M, Plante M, Monchik K, Fleming B, Fadale P. The use of a non-benzodiazepine hypnotic sleep-aid (Zolpidem) in patients undergoing ACL reconstruction: a randomized controlled clinical trial. Knee Surg Sports Traumatol Arthrosc. 2011 May;19(5):787-91. doi: 10.1007/s00167-010-1368-x. Epub 2011 Jan 21. PMID 21253706
- [Background] Wang PK, Cao J, Wang H, Liang L, Zhang J, Lutz BM, Shieh KR, Bekker A, Tao YX. Short-Term Sleep Disturbance-Induced Stress Does not Affect Basal Pain Perception, but Does Delay Postsurgical Pain Recovery. J Pain. 2015 Nov;16(11):1186-99. doi: 10.1016/j.jpain.2015.07.006. Epub 2015 Sep 3. PMID 26342649
- [Background] Xu X, Wang L, Chen L, Su T, Zhang Y, Wang T, Ma W, Yang F, Zhai W, Xie Y, Li D, Chen Q, Fu X, Ma Y, Zhang Y. Effects of chronic sleep deprivation on bone mass and bone metabolism in rats. J Orthop Surg Res. 2016 Aug 2;11(1):87. doi: 10.1186/s13018-016-0418-6. PMID 27485745